CLINICAL TRIAL: NCT00034476
Title: A Phase IIb Study to Determine the Efficacy and Safety of the Study Drug in Patients With Severe Sepsis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1641; J4A-MC-EZZI
Record Dates: First submitted 2002-04-29; First posted 2002-04-30 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Sepsis
Keywords: Sepsis, sPLA2 Inhibitor
MeSH Terms: conditions — Sepsis

INTERVENTIONS:
Drug: sPLA2 Inhibitor

SUMMARY:
The purpose of this study is to determine whether the administration of the study drug is effective in increasing the chance of survival in patients with severe sepsis. Patients entered into this study will be randomly assigned to one of two treatment groups. Patients in each treatment group will be given either the study drug or placebo as a continuous infusion directly into the bloodstream through a catheter placed in one of the patient's veins.

The study drug is an investigational drug that is still in development. It has been studied in approximately 30 healthy subjects, approximately 30 patients with either kidney failure or arthritis, and approximately 600 patients with severe sepsis. Patient participation in this study will last for about one month.

ELIGIBILITY:
Inclusion Criteria: Patients must

* show evidence of acute infection
* meet specified time windows
* be 18 years of age or older

Exclusion Criteria: Patients must not

* have low white blood cell count
* have undergone certain organ transplants
* be HIV positive
* be pregnant or breast feeding
* have severe underlying medical problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466
Dates: Start 2001-10; Study Completion 2002-10

CONTACTS AND LOCATIONS:
Locations (85):
- United States (60):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Berkeley, California
  - Los Angeles, California
  - Orange, California
  - San Diego, California
  - Torrance, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Brandon, Florida
  - Clearwater, Florida
  - Lakeland, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - Oak Park, Illinois
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Lake Charles, Louisiana
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Portland, Maine
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Saint Lous, Missouri
  - Reno, Nevada
  - East Orange, New Jersey
  - New Brunswick, New Jersey
  - Great Neck, New York
  - Manhasset, New York
  - New Hyde Park, New York
  - New York, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Greensboro, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Memphis, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Falls Church, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Belgium (5):
  - Brussels
  - Ghent
  - Liège
  - Ottignies
  - Yvior
- Hungary (7):
  - Budapest
  - Debrecen
  - Debrecend
  - Miskolc
  - Pécs
  - Szeged
  - Vác
- Netherlands (6):
  - 's-Hertogenbosch
  - Apeldoorn
  - Breda
  - Groningen
  - Nijmegen
  - Rotterdam
- Poland (7):
  - Gdansk
  - Krakow-Nowa Huta
  - Poznan
  - Sosnowiec
  - Szczecin
  - Warsaw
  - Wroclaw